CLINICAL TRIAL: NCT06195722
Title: Karadeniz Technical University, Faculty of Health Sciences
Brief Title: Developing a Simulation for Parenteral Drug Administration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sule BIYIK BAYRAM, Karadeniz Technical University, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaradenizTU-2
Record Dates: First submitted 2023-12-12; First posted 2024-01-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Nursing Education; Cognitive Orientation; Injection Site
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): control
- experimental (Experimental): experimental
  Interventions: Other: simulation

INTERVENTIONS:
Other: simulation — parenteral drug simulation
  Arms: experimental

SUMMARY:
In the current Covid-19 pandemic process, distance education has become widespread and will continue to become widespread in the return to normal. In the distance education process, theoretical courses can be given with methods such as synchronous or asynchronous lectures, questions and answers, and discussion. However, in departments such as the nursing department, where laboratory and clinical practice are given during the term, there are some difficulties in providing the practice with distance education. Since students cannot be in clinical practice, they cannot develop their basic nursing skills. However, it is not possible for students to develop their skills in distance education. In addition, due to the high number of students in face-to-face teaching and the low number of lecturers, the lecturer and students cannot spend enough and effective time in the laboratories. Because there are 50-60 students per lecturer and therefore students are not sufficient in basic nursing skills. In order for students to improve their skills, there are technological methods that allow students to try the application on their own, at the desired place and time, without risking patient safety, in virtual environments, without entering the laboratory. Simulation opportunities can be provided to students by creating environments, models, materials and patients similar to the real hospital environment in virtual environments. It is seen in the literature that similar studies have been carried out outside of our country and are used in nursing education. However, in our country, a similar application was made in the virtual environment only in the thesis study of the director. This thesis study, which is similar to this project study, only includes tracheostomy care skill, which is one of the basic nursing skills. This project will include simulation parenteral drug administration skills in our work. For this reason, it will be the first simulation prepared for parenteral drug applications in our country. Drug administration constitutes an important step in patient safety. Although this section is explained theoretically, students are not given sufficient opportunities to have different drug doses prepared and administered in the laboratory. For this reason, when the student encounters a complex situation in the clinic, the decision-making process is prolonged and the risk of making mistakes increases.

DETAILED DESCRIPTION:
In this project study, it is aimed to determine the effect of simulation and teaching to be developed on the knowledge and skills of nursing students in drug administration. For this purpose, a scenario will be written for subcutaneous, intramuscular and intravenous drug administration skills and a simulation will be developed by simulating it in a virtual environment. After the students who accept to participate in the study, take the pre-test and OSCE exam on the subject, the experimental group students will administer the drugs on the virtual patient. After the students they use simulation, a notification will be sent to the researcher's mail address. Thus, it will be determined how many times the students use simulation. When the three-week probation period is over, students will be taken to the posttest and OSCE exam again. Control group students will only follow the laboratory trainings included in the traditional learning process

ELIGIBILITY:
Inclusion Criteria:

* Those who have registered for the Fundamentals of Nursing II Course for the first time,
* Having a computer, tablet or smartphone,
* Having internet access,
* Volunteer to participate in the research

Exclusion Criteria:

* Having graduated from Health Vocational High School or studied a health-related department,
* Have any previous experience of basic nursing skills

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-08-10 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Teaching parenteral drug administration through simulation has an effect on the knowledge test average score of nursing students. | 3 mounth
  Data will be collected through student identification characteristics form, Parenteral Drug Applications Knowledge Test.

SECONDARY OUTCOMES:
Teaching parenteral drug administration through simulation has an effect on the OSCE skill score average of nursing students. | 3 mounth
  Data will be collected through Drug Applications Skill Checklists

CONTACTS AND LOCATIONS:
Overall Officials: Şule Bıyık Bayram, Study Director — Karadeniz Technical University
Locations (1):
- Sule Biyik Bayram, Trabzon, Ortahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No